CLINICAL TRIAL: NCT01572389
Title: Behavioral Activation Therapy for Rural Veterans With Diabetes and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 10-135
Record Dates: First submitted 2012-03-07; First posted 2012-04-06 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus; Depression
Keywords: Diabetes Mellitus; Depression; Affective Symptoms; Self Care; Telemedicine; Psychotherapy
MeSH Terms: conditions — Diabetes Mellitus; Depression; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: HOPE (Experimental): The Healthy Outcomes through Patient Empowerment (HOPE) intervention group is the intervention arm which will employ behavioral health coaching telephone sessions. Tele-coaching is a theoretically grounded, structured processes guided by intervention manuals.
  Interventions: Behavioral: Healthy Outcomes through Patient Empowerment (HOPE)
- Arm 2: EUC (Active Comparator): The Enhanced Usual Care (EUC) group will serve as a concurrent control group to compare to the intervention arm of the study. Participants are screened for diabetes self-management behaviors and control and for active depressive and anxiety symptoms. Primary care providers are alerted of the patients' status and given decision support to enhance care for these uncontrolled conditions.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Healthy Outcomes through Patient Empowerment (HOPE) — HOPE participants will receive 6 behavioral coaching telephone sessions and 3 booster sessions over a six month period followed by usual primary care during the subsequent 6 months maintenance period.
  Arms: Arm 1: HOPE
Behavioral: Enhanced Usual Care — All participants receive usual VA primary care plus a dedicated screening for diabetes control and clinically significant depressive symptoms. Patients and primary care providers are notified of these results and given recommendations for usual care.
  Arms: Arm 2: EUC

SUMMARY:
This clinical trial will compare the effectiveness of the Healthy Outcomes through Patient Empowerment (HOPE) intervention to enhanced usual care (EUC) for diabetes and depression at 6 and 12 month follow-up. The proposed study is a randomized controlled trial enrolling 242 largely rural Veterans with uncontrolled diabetes and clinically-significant depressive symptoms. Both groups will receive screening, education, and notification of clinical findings along with follow-up in usual primary care. HOPE participants will also receive behavioral coaching telephone sessions over a six month period. Patients in the control group will be screened, and providers will be notified of high risk patients' status and need for intervention. Both groups will receive only usual primary care during the subsequent 6 month maintenance period. Study measurements using self-report questionnaires will also be collected at baseline, 6 and 12 months follow-up. The investigators will also conduct chart reviews to evaluate usual care blood tests for diabetes control. Changes in measurements from baseline will be compared between groups. This intervention will reach Veterans in rural setting where community-based primary care is needed, especially care that blends treatment strategies for physical and emotional health.

DETAILED DESCRIPTION:
Project Background: The co-occurrence of diabetes and depressive symptoms is highly prevalent and has dramatic consequences on the quality of life and health of affected patients. Due to the complex interrelation between these conditions, patients often experience both psychological and physiological difficulties. Furthermore, Veterans with diabetes and depressive symptoms in rural settings have limited access to care. Interventions that reach Veterans in rural / community-based primary care are needed, especially those that blend treatment strategies for physical and emotional health.

Project Objectives: Specific (Primary) Aim (1): Compare the effectiveness of the Healthy Outcomes through Patient Empowerment (HOPE) intervention to enhanced usual care (EUC) at 6 and 12 month follow-up.

Hypothesis 1a: After 6 months (active treatment phase), HOPE will produce greater improvements in diabetes control (measured by hemoglobin A1c levels) and depression (measured by PHQ-9 scores) than will EUC.

Hypothesis 1b: At 12 months (6-month active phase plus 6-month maintenance phase), HOPE participants will continue to evidence significant greater improvements in HbA1c and PHQ-9 compared with EUC participants.

Exploratory Specific Aim (2): To examine the role of moderators and mediators on intervention effectiveness Exploratory Aim 2a. To evaluate factors that mediate or moderate effectiveness at 6 and 12 months for all enrolled patients (regardless of intervention group assignment). Potential mediating and moderating variables include patient-level (clinical factors-diabetes distress and self-efficacy and sociodemographics) and facility-level factors (availability of medical and mental health services by clinical site).

Exploratory Aim 2b. To evaluate factors that mediate or moderate effectiveness at 6 and 12 months for patients enrolled in the HOPE intervention arm. Intervention factors include adherence (e.g. session attendance), fidelity (ratings of coach effectiveness), and treatment implementation (e.g., goal setting quality and self-management behaviors) as well as any significant predictors obtained from Aim 1a.

Exploratory Specific Aim (3): Evaluate the potential for embedding the HOPE intervention processes within a VA CBOC using the REAIM framework for evaluating effectiveness of behavioral interventions.

Exploratory Aim 3a - Reach. Compare clinical and demographic characteristics of enrolled study participants with the characteristics of all potentially eligible patients at each CBOC.

Exploratory Aim 3b - Adoption. Qualitatively elicit clinicians' perceptions of behavioral coaches, patients' use of action plans, and responses to coaches' recommendations in preparation for future implementation

Project Methods: The proposed study is a randomized controlled trial enrolling 242 largely rural Veterans with uncontrolled diabetes and clinically-significant depressive symptoms. Both groups will receive screening, education, and notification of clinical findings along with follow-up in usual primary care. HOPE participants will also receive 6 behavioral coaching telephone sessions and 3 booster sessions over a six month period. Coaches will use a standardized, theory-based process for conducting the sessions with the aim of creating patient-centered and articulated goals and behavioral action plans. Participants' primary care providers will be notified about session discussions and the resultant goals and action plans. Both groups will receive only usual primary care during the subsequent 6 months maintenance period. Hemoglobin A1c and PHQ-9 measurements along with self-report questionnaires will also be collected at baseline, 6 and 12 months follow-up. Changes in measurements from baseline will be compared between groups. Analytic evaluations of intervention mediators/moderators and implementation will also be conducted at 6 and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with comorbid diabetes and depressive symptoms receiving primary care services at VA CBOCs throughout Southeast Texas
* as well as MEDVAMC patients living >20 miles from the hospital who face similar distance related treatment barriers

Participants must have:

* a diagnosis of diabetes mellitus
* an average HbA1c level >7.5% in the prior 6 months
* clinically significant symptoms of depression
* Verification of diabetes mellitus diagnoses will be based on data collected from the VA data warehouse.
* To verify that participants meet the depression criteria, the investigators will use participant self-report of clinically significant depressive symptoms according to the PHQ-9, where a score of greater than/equal to 10 on the PHQ-9 will signify a clinically meaningful symptom burden.

Exclusion Criteria:

* The investigators will exclude potential participants only for clinical factors that would render a telephone-based behavioral activation intervention inappropriate.
* Specific exclusion criteria are:

  * lack of regular access to a telephone
  * significant cognitive impairment (three or more errors) on an established six-item screening exam
  * meeting criteria for bipolar, psychotic, or substance-abuse disorders
  * presence of uncorrected hearing or vision impairment
  * their medical chart recommends not titrating therapy due to prior history of significant hypoglycemic events
  * they live within 20 miles of the MEDVAMC.
* Patients will be secondarily excluded if their HbA1C level falls below 7.5% at baseline assessment, or if they report suicidal ideation on the PHQ-9 at baseline assessment.
* Patients receiving mental health services at the time of study recruitment will not be excluded.
* All mental health treatments and health service-use characteristics will be included in study analyses as covariates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aanand D Naik, MD BA, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX; Jeffrey Cully, PhD MEd, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin CE, Renn BN, Winderman KE, Hundt N, Petersen NJ, Naik AD, Cully JA. Classifying diabetes-burden: A factor analysis of the Problem Areas in Diabetes Scale. J Health Psychol. 2018 May;23(6):882-888. doi: 10.1177/1359105316678667. Epub 2016 Nov 21. PMID 27872390
- [Result] Tinetti ME, Naik AD, Dodson JA. Moving From Disease-Centered to Patient Goals-Directed Care for Patients With Multiple Chronic Conditions: Patient Value-Based Care. JAMA Cardiol. 2016 Apr 1;1(1):9-10. doi: 10.1001/jamacardio.2015.0248. No abstract available. PMID 27437646
- [Result] Naik AD, Lawrence B, Kiefer L, Ramos K, Utech A, Masozera N, Rao R, Petersen NJ, Kunik ME, Cully JA. Building a primary care/research partnership: lessons learned from a telehealth intervention for diabetes and depression. Fam Pract. 2015 Apr;32(2):216-23. doi: 10.1093/fampra/cmu084. Epub 2014 Dec 31. PMID 25552674
- [Result] Cully JA, Breland JY, Robertson S, Utech AE, Hundt N, Kunik ME, Petersen NJ, Masozera N, Rao R, Naik AD. Behavioral health coaching for rural veterans with diabetes and depression: a patient randomized effectiveness implementation trial. BMC Health Serv Res. 2014 Apr 28;14:191. doi: 10.1186/1472-6963-14-191. PMID 24774351
- [Result] Naik AD, White CD, Robertson SM, Armento ME, Lawrence B, Stelljes LA, Cully JA. Behavioral health coaching for rural-living older adults with diabetes and depression: an open pilot of the HOPE Study. BMC Geriatr. 2012 Jul 24;12:37. doi: 10.1186/1471-2318-12-37. PMID 22828177
- [Derived] Vaughan EM, Cully JA, Petersen NJ, Hundt NE, Kunik ME, Zeno DD, Naik AD. Testing the Impact of a Collaborative, Goal-Setting, and Behavioral Telehealth Intervention on Diabetes Distress: A Randomized Clinical Trial. Telemed J E Health. 2022 Jan;28(1):84-92. doi: 10.1089/tmj.2020.0533. Epub 2021 Mar 15. PMID 33728989
- [Derived] Naik AD, Hundt NE, Vaughan EM, Petersen NJ, Zeno D, Kunik ME, Cully JA. Effect of Telephone-Delivered Collaborative Goal Setting and Behavioral Activation vs Enhanced Usual Care for Depression Among Adults With Uncontrolled Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e198634. doi: 10.1001/jamanetworkopen.2019.8634. PMID 31390035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 225 participants enrolled into the study. Consent occurred at baseline and participants were eligible if they scored a 10 or greater on the PHQ-9 and an A1C of 7.5 or greater. If a participant didn't meet these criteria then they were not randomized into the study.
Period: Overall Study
Arm/Group | Arm 1: HOPE | Arm 2: EUC
Started | 136 | 89
Completed | 90 | 68
Not Completed | 46 | 21
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 14 | 2
Not completed — Lost to Follow-up | 25 | 14
Not completed — Only A1C or Assessment was Collected | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: HOPE | Arm 2: EUC | Total
Number analyzed (Participants) | 136 | 89 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.4) | 60.8 (8.0) | 61.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 121 | 81 | 202
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 73 | 51 | 124
  Race: Black | 41 | 16 | 57
  Race: Hispanic | 12 | 11 | 23
  Race: Other | 2 | 4 | 6
  Race: More than 1 race | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1C
Description: Measures of Hemoglobin A1C will be taken to assess average blood glucose levels throughout the study as an indicator of diabetes control. Hemoglobin A1C is a blood test taken to assess average blood glucose levels in the body. Normal range of A1C level is below 5.7. Eligible participants had an A1C of 7.5 or higher. The higher the A1C the more a person's diabetes is uncontrolled.
Time Frame: Hemoglobin A1C levels will be measured at baseline, 6-, and 12- months.
Population: The number analyzed at each timepoint decreased due to non-completion of the A1C blood draw by participants.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Arm 1: HOPE | Arm 2: EUC
Number analyzed (Participants) | 136 | 89
percentage of glycated hemoglobin
  Baseline | 9.2 (1.4) | 9.3 (1.5)
  6-Months: number analyzed (Participants) | 105 | 78
  6-Months | 9.1 (1.7) | 8.7 (1.7)
  12-Months: number analyzed (Participants) | 90 | 68
  12-Months | 8.7 (1.6) | 8.9 (2)

2. Primary Outcome: Change in Patient Health Questionnaires-9 During Intervention
Description: The Patient Health Questionnaires-9 assesses depressive symptoms during the course of the intervention. The PHQ-9 ranges in score from 0 - 27; where higher numbers represent increase levels of depression. Scores from 5 - 9 represent "minimal symptoms" of depression; 10 - 14 represent "minor depression", dysthymia, or major depression - mild; 15 - 19 represent "major depression, moderately severe"; and scores of 20 and above is considered "major depression, severe." Participants with that scored a 10 or above were eligible for the study.
Time Frame: PHQ-9 will be assessed at baseline, 6-, and 12- months.
Population: The number analyzed at each timepoint decreased due to non-completion of the assessment by participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: HOPE | Arm 2: EUC
Number analyzed (Participants) | 136 | 89
units on a scale
  baseline | 15.8 (4.2) | 16.2 (4)
  6 Months: number analyzed (Participants) | 105 | 78
  6 Months | 10.9 (6.1) | 12.4 (6)
  12 Months: number analyzed (Participants) | 90 | 68
  12 Months | 10.1 (6.9) | 12.6 (6.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 6 and 12 months at the time of assessments.
Arm/Group | Arm 1: HOPE | Arm 2: EUC
All-Cause Mortality (participants affected / at risk) | 1/136 | 3/89
Serious Adverse Events (participants affected / at risk) | 1/136 | 0/89
Other Adverse Events (participants affected / at risk) | 0/136 | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: HOPE (N=136) | Arm 2: EUC (N=89)
Foot Sore (Infections and infestations) | 1 (1) | 0 (0) — Patient indicated to his coach he had a sore on his foot that would not heal. He followed up with his physician and there was concern about the length of time it was taking to heal. There was no indication the sore was due to his participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No